CLINICAL TRIAL: NCT04697355
Title: Case Study to Evaluate the Safety and Effect on Energy Expenditure of Naringenin and Beta Carotene
Brief Title: Effect of Naringenin and Beta Carotene on Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Chief Medical Officer, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB FWA 00006218
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-04

CONDITIONS: Energy Expenditure; Safety Issues; Glucose Metabolism
MeSH Terms: interventions — naringenin; beta Carotene

STUDY DESIGN:
Intervention Model Description: Case study in a single human subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Naringenin + Beta carotene (Experimental): Subject will ingest 300 mg naringenin three times/day and 6 mg beta carotene two times/day
  Interventions: Dietary Supplement: naringenin and beta carotene

INTERVENTIONS:
Dietary Supplement: naringenin and beta carotene — Subject will ingest 300 mg naringenin three times/day and 6 mg beta carotene two times/day for eight weeks

SUMMARY:
This study is designed to test the effects of the combination of naringenin (from an extract of sweet oranges) and beta carotene on energy expenditure and glucose metabolism in a single human subject.

DETAILED DESCRIPTION:
The subject will be treated for 8 weeks with the combination of naringenin + beta carotene.

We will conduct the following assessments before the treatment and at the end of eight weeks.

1. Resting metabolic rate
2. Oral glucose tolerance test with glucose and insulin
3. Ambulatory blood pressure
4. Recording of adverse events
5. Body weight

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose < 200mg/dL

Exclusion Criteria:

* Known allergy to citrus fruits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | Five hours
  Ventilated hood
Incidence of Treatment-Emergent Adverse Events | Eight weeks
  Adverse events

SECONDARY OUTCOMES:
Glucose metabolism | Three hours
  Oral glucose tolerance test with insulin
Blood pressure | 24 hours
  Ambulatory
Body weight | 16 weeks
  Measurement of body weight

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Greenway, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murugesan N, Woodard K, Ramaraju R, Greenway FL, Coulter AA, Rebello CJ. Naringenin Increases Insulin Sensitivity and Metabolic Rate: A Case Study. J Med Food. 2020 Mar;23(3):343-348. doi: 10.1089/jmf.2019.0216. Epub 2019 Oct 31. PMID 31670603